CLINICAL TRIAL: NCT00381784
Title: Connect-To-Protect® Phase III: Local Evaluation of Community Promise Connect-To-Protect® Phase III: Local Evaluation of Mpowerment
Brief Title: C2P - Phase III: MPowerment and Community Promise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ATN 041
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2016-03

CONDITIONS: HIV Infections
Keywords: YMSM; HIV/AIDS; Condom use; Drug users; Minority women
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Drug Misuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Community PROMISE (Experimental): Community PROMISE is a community level HIV/STD prevention program that relies on role model stories and peer advocates from the community. Sites will adapt PROMISE for local use remaining faithful to the core elements.
  Interventions: Behavioral: Printed materials
- Mpowerment (Experimental): MPowerment is a community level HIV/STD prevention program that relies on peer advocates from the community to lead outreach activities including discussion groups (Mgroups), venue-based outreach, social events and a publicity campaign. Sites will adapt MPowerment for local use remaining faithful to the core elements.
  Interventions: Behavioral: Peer advocates

INTERVENTIONS:
Behavioral: Printed materials — Role model stories comprise the "heart" of printed materials distributed throughout the target community. The role model stories are brief publications that depict personal accounts from individuals in the population of focus who have made or are planning to make a risk-reducing behavioral change. Depending on the population they are meant to reach and what behavior they are trying to influence, the stories may include examples of people who now carry condoms with them, talked to a partner about condom use, use condoms consistently, avoid sharing needles, or exhibited other risk reduction behaviors.
  Other Names: No other names.
  Arms: Community PROMISE
Behavioral: Peer advocates — Core Element 1 Core group of young gay men and additional volunteers recruited from the community. The core group and volunteers comprise the "peer advocates" who design and carry out all program activities.
  Core Element 2 Designated space where most social events and meetings are held; also serves as a drop in center where young men can meet and socialize during specified hours.
  Core Element 3 Social events to attract young gay men and to promote safer sex. Core Element 4 Teams of young gay men go to locations frequented by young gay men to discuss and promote safer sex, deliver appealing informational literature on HIV risk reduction and distribute condoms.
  Core Element 5 Meetings of eight to 10 young gay men to discuss factors contributing to unsafe sex among men. Men practice safer sex negotiation and correct condom use skills.
  Core Element 6 Publicity campaigns that attract men to the program by word of mouth and through articles and advertisements in gay newspapers.
  Other Names: There are no other names.
  Arms: Mpowerment

SUMMARY:
One of the objectives of the C2P coalition is the successful delivery of a CDC-endorsed community-level HIV prevention program aimed at changing the risk profiles of youth. This protocol (ATN 041) describes the program, Community PROMISE (Peers Reaching Out and Modeling Intervention Strategies) or MPowerment, and plans for adapting and implementing it. There are a total of 4 interventions that a community can implement.

DETAILED DESCRIPTION:
Community Promise: Role model stories comprise the "heart" of printed materials distributed throughout the target community. The role model stories are brief publications that depict personal accounts from individuals in the population of focus who have made or are planning to make a risk-reducing behavioral change. The messages in the role model stories are reinforced by interpersonal communication with trained peer advocates.

MPowerment: is a community level HIV/STD prevention program that relies on peer advocates from the community to lead outreach activities including discussion groups (M-groups), venue-based outreach, social events and a publicity campaign. Sites will adapt MPowerment for local use remaining faithful to the core elements.

ELIGIBILITY:
Community Promise:

Inclusion Criteria

1. Adolescents and young adults who provide verbal confirmation that their age is within
2. the range of 12 through 24 years, inclusive.
3. Gender will reflect that of the population of focus.
4. Must report having engaged in voluntary sexual activity within the past 12 months (vaginal, anal and/or oral sex).
5. Ability to understand and willingness to provide informed consent/assent.

Exclusion Criteria

1. Visibly distraught and/or visibly emotionally unstable (e.g., depressive mood, or exhibiting manic, suicidal, or violent behavior).
2. Visibly intoxicated or under the influence of psychoactive agents
3. Clinically presents as acutely ill.

MPowerment:

Inclusion Criteria

1. Male adolescents and young adults who provide verbal confirmation that their age is within the range of 12 through 24 years, inclusive.
2. Must report having engaged in voluntary sexual activity within the past 12 months (anal and/or oral sex) with a man.
3. Ability to understand and willingness to provide informed consent/assent.

Exclusion Criteria

1. Visibly distraught and/or visibly emotionally unstable (i.e., depressive mood,
2. or exhibiting manic, suicidal, or violent behavior, etc.).
3. Visibly intoxicated or under the influence of psychoactive agents.
4. Clinically presents as acutely ill.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2006-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The goal of PROMISE and Mpowerment is to effect community change through diffusion of health-promoting information via naturally occurring social networks. Data collection is process evaluation data only. | 4 years

SECONDARY OUTCOMES:
Successful delivery of a CDC-endorsed community-level HIV prevention program | 4 years
  One of the objectives of the C2P coalition is the successful delivery of a CDC-endorsed community-level HIV prevention program aimed at changing the risk profiles of youth.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ellen, MD, Study Chair — Johns Hopkins University
Locations (7):
- United States (6):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Childrens Hospital National Medical Center, Washington D.C., District of Columbia
  - USF Peds Division of Infectious Disease, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
- University Pediatric Hospital, San Juan, Puerto Rico

REFERENCES:
- See also: ATN website — http://www.atnonline.org